CLINICAL TRIAL: NCT05787912
Title: Efficacy of Hyaluronic Acid Gel and Photobiomodulation on Wound Healing After Surgical Gingivectomy: a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Hyaluronic Acid Gel and Photobiomodulation on Wound Healing After Surgical Gingivectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Basma Khalil, Resident of Periodontology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #1
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Gingival Enlargement
Keywords: Surgical gingivectomy; Hyaluronic acid; Photobiomodulation
MeSH Terms: conditions — Gingival Hyperplasia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation (Experimental)
  Interventions: Device: Photobiomodulation
- Hyaluronic acid gel after photobiomodulation (Experimental)
  Interventions: Other: Hyaluronic acid after photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — The surgical sites were irradiated with a diode laser (980 nm, 0.2W) only.
  Arms: Photobiomodulation
Other: Hyaluronic acid after photobiomodulation — The surgical sites after gingivectomy were irradiated with a diode laser (980 nm, 0.2W) then covered by 2% Hyaluronic acid gel loaded in a special appliance for each patient.
  Arms: Hyaluronic acid gel after photobiomodulation

SUMMARY:
The aim of this study was to evaluate the effect of hyaluronic acid gel after photobiomodulation on the healing of surgical gingivectomy sites

ELIGIBILITY:
Inclusion Criteria:

* Chronic inflammatory gingival enlargement grade 2 and 3 according to the gingival overgrowth index by Miller and Damn.
* Adequate amount of keratinized tissue.
* Attachment loss= 0
* Well educated patients as post-operative instructions need to be followed precisely.

Exclusion Criteria:

* Patients with history of smoking
* Pregnant women
* Patients with bad oral hygiene
* Patients who have any known systemic disease that interfere with performance of surgical gingivectomy or periodontal wound healing
* Patients who have any previous adverse reactions to the products (or similar products) used in this study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Wound healing | up to 21 days
  Assessed using Landry's healing index which grades the wound on a scale of 1 (poor) to 5 (excellent)
  * Very poor (1): ≥50% of gingiva red, bleeding on palpation, Granulation tissue present, Non-epithelialized incision margin with loss of epithelium beyond the margin.
  * Poor (2): ≥50% of gingiva red, bleeding on palpation, Granulation tissue present, Non-epithelialized incision margin with exposed connective tissue
  * Good (3): ≥25% and<50% of gingiva red, No bleeding on palpation, no granulation tissue, No exposed connective tissue on the incision margin
  * Very good (4): <25% of gingiva red, No bleeding on palpation, no granulation tissue, No exposed connective tissue on the incision margin
  * Excellent (5): All tissues are pink, No bleeding on palpation, no granulation tissue, No exposed connective tissue on the incision margin
Perceived pain | up to 21 days
  This was assessed using Visual Analogue Scale (VAS). Patients were instructed to chart their perceptions of pain using VAS ranging from 0-10; where 0 represents no pain/burning sensation and 10 represents severe pain/burning sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Basma K Yacout, BDS, Principal Investigator — Alexandria University; Fatma R Kamel, PhD, Study Director — Alexandria University; Maha A Abou Khadr, PhD, Study Director — Alexandria University; Lamia A Heikal, PhD, Study Director — Faculty of Pharmacy, Alexandria University; Gillan I El-Kimary, PhD, Study Chair — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Yakout BK, Kamel FR, Khadr MAEA, Heikal LAH, El-Kimary GI. Efficacy of hyaluronic acid gel and photobiomodulation therapy on wound healing after surgical gingivectomy: a randomized controlled clinical trial. BMC Oral Health. 2023 Oct 27;23(1):805. doi: 10.1186/s12903-023-03519-5. PMID 37891549